CLINICAL TRIAL: NCT05234411
Title: Ketonemia Through Menstrual Cycle
Acronym: KETOMENS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Collaborators: IRCCS ISTITUTO NEUROLOGICO CASIMIRO MONDINO (Unknown)
Responsible Party: Principal Investigator, Cinzia Ferraris, Researcher, University of Pavia
Other Study IDs: 2021-KETOMENS
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy; Drug Resistant Epilepsy; GLUT1DS1; Ketogenic Dieting; Menstrual Epilepsy
Keywords: ketogenic diet; ketonemia; menstrual cycle
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy; Ketosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Eligible participants will be female patients aged 13 years or older, with regular menstrual cycle, who have been undergoing a KDT for at least 3 months and thus previously diagnosed with Drug resistant epilepsy or GLUT1DS.
  Interventions: Other: Evaluation of ketogenic diet impact on ketonemia

INTERVENTIONS:
Other: Evaluation of ketogenic diet impact on ketonemia — Ketonemia and glycemia levels monitoring during different phases of menstrual cycles

SUMMARY:
Ketogenic dietary therapies (KDTs) are well-established, safe, non-pharmacologic treatments used for children and adults with drug-resistant epilepsy and other neurological disorders. Ketone bodies levels undergo a significant inter-individual and intra-individual variability and can be affected by several factors. This evidence suggests the need for personalized monitoring for diet optimization, especially at the beginning of the treatment but during whole follow-up. Possible variations in glycemia and ketone bodies' blood level according to different phases of menstrual cycle have not been systematically assessed yet, but this time window deserves special attention because of hormonal and metabolic related changes. We present the methodological protocol for a longitudinal, multicentric study aimed at searching for subtle changes in ketone bodies blood level during menstrual cycle in epileptic female patients undergoing a stable ketogenic diet. The study will be divided into two phases. The first one will be purely observational, aiming at the assessment of ketonemia during menstrual cycle. Whether this finding will be confirmed, a second phase of ketogenic diet therapy adjustment will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with drug resistant epilepsy or GLUT1DS undergoing KD from at least 3 months before inclusion to the study
* Patients who had menarche at least 3 months before inclusion to the study
* Absence of recognized endocrinologic problems/ disease

Exclusion Criteria:

* Patients who experienced secondary amenorrhea
* Patients who have irregular menstrual cycle
* Pregnant patients

Ages: 12 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — * Patients who had menarche at least 3 months before inclusion to the study
  * Patients undergoing KDTs from at least 3 months
Study Population: Eligible participants will be female patients aged 13 years or older, with regular menstrual cycle, who have been undergoing a KDT for at least 3 months and thus previously diagnosed with Drug resistant epilepsy or GLUT1DS.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To measure serum ketone bodies level through different phases of menstrual cycle | 3 months
  With regular home standardized measurements of capillary ketonemia

SECONDARY OUTCOMES:
Evaluation of the efficacy of an individualized intermittent adjustment of the dietary regimen | 3 months
  Evaluation of ketonemia levels and clinical outcome once the therapeutic intervention is implemented

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasca L, Ferraris C, Guglielmetti M, Varesio C, Totaro M, Trentani C, Marazzi C, Brambilla I, Ballante E, Armeno M, Valenzuela GR, Caraballo RH, Veggiotti P, Tagliabue A, De Giorgis V. Ketonemia variability through menstrual cycle in patients undergoing classic ketogenic diet. Front Nutr. 2023 Jul 27;10:1188055. doi: 10.3389/fnut.2023.1188055. eCollection 2023. PMID 37575326